CLINICAL TRIAL: NCT04729790
Title: Phase II Randomized Clinical Trial of Standard FMT Treatments: Non-powered Pilot Study of the Safety and Efficacy of Orally Administered Lyophilized Fecal Microbiota Product (PRIM-DJ2727) for the Treatment of Recurrent Clostridium Difficile Infection (RCDI) Using Either Single or Three Combined Products From Healthy Donors
Brief Title: Randomized Clinical Trial of Standard FMT Treatments
Acronym: FMT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Herbert DuPont, MD, Professor of Infectious Diseases, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-SPH-19-0950
Record Dates: First submitted 2021-01-20; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Clostridium Difficile

STUDY DESIGN:
Intervention Model Description: This is a double-blinded study for the groups randomized to receive FMT products either from single or three healthy donors
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent statistician will develop a randomization list using SAS. Randomization in permuted blocks will be used to achieve balance across treatment groups. The randomization scheme consists of a sequence of blocks such that each block contains a pre-specified number of treatment assignments in random order. The purpose of this is to balance the randomization scheme at the completion of each block. The target sample size is 200 evaluable subjects or as many as can be done up to that number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with RCDI will receive FMT capsules from single donor (Active Comparator): Capsules made with intestinal bacteria from single healthy donor
  1. st treatment day, lyophilized product generated from single donor (90g of stool)
  2. nd treatment day, lyophilized product generated from single donor (90g of stool)
  Interventions: Drug: PRIM-DJ2727
- Patient will receive FMT capsules from three donors (Experimental): Capsules made of intestinal bacteria from three healthy donors
  1. st treatment day, lyophilized product generated from three donors (90g of stool)
  2. nd treatment day, lyophilized product generated from three donors (90g of stool)
  Interventions: Drug: PRIM-DJ2727

INTERVENTIONS:
Drug: PRIM-DJ2727 — oral FMT capsules

SUMMARY:
This is a single center, randomized, parallel assignment, double-blinded, efficacy and safety study to be conducted in subjects with recurrent C. difficile Infection (RCDI). Approximately 200 subjects will be enrolled in the study and randomized at 1:1 ratio to receive lyophilized intestinal bacteria obtained from either single or three donors (group 1 receiving healthy microbiota collected from single donor 90g stool for 2 consecutive days; group 2 receiving healthy microbiota collected from three donors 90g stool for 2 consecutive days). All subjects will be followed for approximately 180 days following FMT treatment for safety.

DETAILED DESCRIPTION:
The endpoints of the study are to evaluate the efficacy and safety of lyophilized product by capsules obtained either from single or three donors and the prevention of subsequent bouts of CDI in 60 days post FMT.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years of age or older.
2. Sexually active male and female subjects of childbearing potential agree to use an effective method of birth control during the study.
3. Female subjects of childbearing potential will be asked if they could be pregnant. If the subject is unsure a pregnancy test will be completed
4. Subject/LAR willing and able to provide informed consent.
5. Able to follow study procedures and complete the follow-up questionnaire for safety.
6. Subject must have an attending physician who will provide non-transplant care (Either PI of this study or referring physician).
7. Medical history of ≥ 3 bouts of CDI in outpatient or ≥ 2 bouts of CDI in inpatient with either group having ≥ 2 positive fecal tests for C. difficile toxin and at least one bout of CDI within 6 months of enrollment.
8. Received at least two courses of standard-of-care antibiotic therapy for CDI.

Exclusion Criteria:

1. Unable to take capsules orally.
2. Requiring systemic non-C. difficile antibiotic therapy within 14 days prior to FMT.
3. Unwilling to stop taking non-dietary probiotics 24-96 hours prior to FMT.
4. Unable to stop taking bile acid sequestrants (e.g. cholestyramine) 24-96 hours prior to FMT.
5. Unable to stop use of drugs with CDI activity: oral vancomycin, oral or IV metronidazole, fidaxomicin, rifaximin or nitazoxanide 24-96 hours prior to FMT and after FMT.
6. Receipt of CDI monoclonal antibodies as treatment for the most recent bout of CDI.
7. Life expectancy of < 6 months.
8. In the opinion of investigator, subject for any reason, should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of participants with treatment-related adverse events | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Herbert l DuPont, MD, Study Director — University of Texas Health Science Center School of Public Health

IPD SHARING:
Plan to Share IPD: No